CLINICAL TRIAL: NCT02145507
Title: Clinical Investigation to Evaluate the Haemonetics LeukoSep Leukocyte Reduction Filtration System for Whole Blood With CPD Anticoagulant and SOLX Additive - Pivotal Trial
Brief Title: Evaluation of Whole Blood With CPD Anticoagulant and AS-7/SOLX Additive Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: TP-CLN-100331
Record Dates: First submitted 2014-05-19; First posted 2014-05-23 (Estimated); Results first posted 2022-03-28 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Blood Donors
Keywords: Leukoreduction; Red Blood Cell post-leukoreduction recovery; Packed red blood cell post storage hemolysis; Red blood cell recovery; Plasma clotting factors; 2,3-DPG rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Room Temperature Storage/Filtration (Other): SOLX (Investigational Product) and AS-3 (Control)
  Interventions: Drug: SOLX (Investigational); Drug: AS-3 (Control)
- Arm 2 : Cold storage (Other): SOLX (Investigational Product) and AS-3 (Control)
  Interventions: Drug: SOLX (Investigational); Drug: AS-3 (Control)

INTERVENTIONS:
Drug: SOLX (Investigational) — SOLX is regulated as a drug but is not intended to provide a direct therapeutic benefit.
  Other Names: AS-7; Additive solution 7
Drug: AS-3 (Control) — AS-3 solution is regulated as a drug but is not intended to provide a direct therapeutic benefit
  Other Names: Additive solution formula 3

SUMMARY:
This study will evaluate a new blood collection and filtration system that is intended to be used to collect, filter, separate and store red blood cells and, separately, plasma. The new blood collection and filtration system will be compared to an already-approved and currently used system. Further, this study will evaluate new processing conditions relative to the individual components of the collection and filtration system. All study participants will donate two units of whole blood with individual units being donated at least 56 days apart. One unit of whole blood will be donated with the new system, and the other unit will be collected with the already-approved system. A subset of the donors (approximately 24 of the 120 participants) will have a small quantity of their red blood cells injected back into their body 42-days after they were donated in order to evaluate how well the red blood cells survive. Blood and blood products from all donors will be analyzed the day of collection and after storage (plasma after at least 30 days of storage and red blood cells after exactly 42 days of storage).

DETAILED DESCRIPTION:
In vitro and in vivo performance of SOLX® RBCs produced with the modified SOLX® System will be used to demonstrate the acceptability of both the proposed product modification and expanded indications. To accomplish this, the study will require a total of 120 evaluable donors completing the study. Enrolled donors will be assigned to either of two study arms. Each study arm will entail a randomized, paired, 2-x-2 crossover design where every study donor (n = 60 evaluable study donors who complete the study per arm) will donate a total of two whole blood units with individual units being donated at least 56 days (8 weeks) apart. One unit will be collected with the investigational product (IP) and the other unit will be collected with the control product (CP). The order in which the IP and the CP will be used to collect, filter and store the whole blood and appropriate blood products (within the context of the crossover design) will be randomized.

Each of the two study arms will evaluate outcomes resulting from different storage, filtration and processing conditions:

* Arm 1 will entail holding whole blood units at 20-24°C after collection for ≥ 20 hours (IP) or ≥ 6 hours (CP) prior to initiating room temperature filtration. Following room temperature centrifugation and subsequent separation, SOLX® PRBC will be placed at 1-6°C and plasma placed at ≤ -18°C within 24 hours (IP) or within 8 hour (CP) of collection. The first donation will occur with product indicated per randomization and the second donation will occur with product alternate to the randomization. Arm 1 will further entail an in vivo double-radiolabelled autologous RBC recovery substudy (n = 20-24, paired IP and CP data will be collected) and an evaluation of pre- and post-rejuvenation PRBC 2,3-DPG levels (all IP and CP units). The in vivo substudy and rejuvenation evaluation is limited to only Arm 1 and is not included in Arm 2.
* Arm 2 will entail holding whole blood units at 1-6°C after collection for ≥ 66 hours (both IP and CP) prior to initiating cold filtration. Following refrigerated centrifugation and subsequent separation, SOLX® PRBCs will be placed at 1-6°C within 72 hours of collection (both IP and CP). Plasma will not be evaluated for this arm and will be discarded. The first donation will occur with product indicated per randomization and the second donation will occur with product alternate to the randomization.

For each study arm that does not meet the protocol-defined in vitro acceptance criteria for exactly 1 unit, an additional 71 evaluable donors will be enrolled, thus increasing the number of evaluable enrolled donors completing the respective study arm to 131 donors. Only those acceptance criteria endpoints that were not met within their respective study arm will be evaluated and neither matched/paired crossover controls nor in vivo RBC recovery (Arm 1 In vivo substudy) will be evaluated. If all protocol defined in vitro acceptance criteria are met or > 1 subject does not meet the protocol defined in vitro acceptance criteria relative to a specific study arm, then no enrollment will occur relative to the same study arm.

ELIGIBILITY:
Inclusion Criteria:

* Age - Study donor must be ≥ 18 years of age
* Weight - Study donor must be ≥ 110 pounds
* Temperature - Study donor's body temperature must be ≤ 37.5°C / 99.5°F (oral)
* Hemoglobin - Study donor's hemoglobin must be ≥12.5 g/dL
* Hematocrit - Study donor's hematocrit must be ≥ 38%. Donor Eligibility - Study donor must meet all criteria per respective site's Research Blood Donation Record (BDR)
* Prior Donation - Study donor's most recent single RBC unit donation must have been ≥56 days prior to study donation. Study donor's most recent double RBC unit donation must have been ≥ 112 days prior to study donation
* Informed Consent - Study donor must have consented to study participation by reviewing and having expressed understanding the site-respective IRB-approved informed consent form prior to undergoing any study related procedures
* Blood-borne Pathogens - Study donor's testing results from collected blood does not indicate a risk of transfusion-transmitted disease (TTD)
* Adverse Events - Study donors must agree to report adverse events from the time of signing the informed consent to twenty-four hours following the end of their active study involvement
* Pregnancy - Female study donors must not be pregnant, expected to be pregnant or breastfeeding. Only female donors who participate in the in vivo portion of the study: Women of child-bearing age must not be pregnant as determined by a negative pregnancy test prior to each re-infusion. If acceptable by local procedures, post-menopausal or surgically sterile women may be exempt from the pregnancy testing requirement

Exclusion criteria:

-Failure to meet one or more of the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lou A Maes, MD, Principal Investigator — ARC Mid-Atlantic Region Blood Services; Jose Cancelas, MD, Principal Investigator — Hoxworth Blood Center
Locations (2):
- United States (2):
  - Hoxworth Blood Center, Cincinnati, Ohio
  - American Red Cross Mid-Atlantic Region Blood Services, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 170 participants were enrolled. 82 participants were enrolled in Arm 1 and 88 participants were enrolled in Arm 2. In Arm 1, 70 participants successfully completed the first donation, and 63 completed the second donation. In Arm 2, 67 participants successfully completed the first donation, and 60 completed the second donation.
Groups:
- Arm 1: Room Temperature: Whole blood donation for room temperature storage of IP and CP.
  SOLX (Investigational Product): SOLX is regulated as a drug but is not intended to provide a direct therapeutic benefit.
  AS-3 (Control): AS-3 solution is regulated as a drug but is not intended to provide a direct therapeutic benefit.
- Arm 2: Cold Storage: Whole blood donation for cold storage for IP and CP.
  SOLX (Investigational Product): SOLX is regulated as a drug but is not intended to provide a direct therapeutic benefit.
  AS-3 (Control): AS-3 solution is regulated as a drug but is not intended to provide a direct therapeutic benefit.
Period: First Donation
Arm/Group | Arm 1: Room Temperature | Arm 2: Cold Storage
Started | 82 | 88
Randomized to Have Blood Processed With SOLX (IP) | 52 | 51
Randomized to Have Blood Processed With AS-3 (CP) | 30 | 37
Completed | 70 | 67
Not Completed | 12 | 21
Period: Second Donation
Arm/Group | Arm 1: Room Temperature | Arm 2: Cold Storage
Started | 65 | 65 (Note: Of the 65 participants who started the second period in Arm 2, there were 3 screen failures, therefore only n=62 participants received their alternate procedure.)
Blood Processed With AS-3 (CP) | 39 | 35
Blood Processed With SOLX (IP) | 26 | 27
Completed | 63 | 60
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Population: Donors who consented to study participation and who successfully donated blood ≥ 1 time (maximum donations = 2).
Groups:
- Arm 1: Room Temperature Storage/Filtration: In vitro whole blood storage, leukoreduction and processing of donated whole blood.
  SOLX: SOLX is regulated as a drug but is not intended to provide a direct therapeutic benefit.
- Arm 2 : Cold Storage/Filtration: In vitro analysis of whole blood following refrigerated storage for > 66 hours prior to leukoreduction and subsequent processing of packed red blood cells.
  SOLX: SOLX is regulated as a drug but is not intended to provide a direct therapeutic benefit.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Room Temperature Storage/Filtration | Arm 2 : Cold Storage/Filtration | Total
Number analyzed (Participants) | 82 | 88 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (13.05) | 38.7 (14.24) | 41.1 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 46 | 91
  Male | 37 | 42 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 81 | 83 | 164
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 11 | 10 | 21
  White | 69 | 70 | 139
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 82 | 88 | 170

OUTCOME MEASURES:

1. Primary Outcome: Red Blood Cell Post-filtration Recovery
Description: The percent of recovered red blood cells when the content of pre-filtration whole blood is compared to the post-filtration leukoreduced whole blood content.
Time Frame: Arm and product dependent (< 8 hours, 20-24 hours, 66-72 hours post collection)
Population: Population represents matched samples from the same donor (i.e., each donor's blood was collected with the SOLX set and the Control set, and as such, Arm 1 represents 60 donors and Arm 2 represents 58 donors).
Measure: Mean (Standard Deviation); unit: % recovery at day 0
Groups:
- Arm 1: SOLX Room Temperature Storage/Filtration: SOLX (Investigational Product)
  SOLX (Investigational): SOLX is regulated as a drug but is not intended to provide a direct therapeutic benefit.
  AS-3 (Control): AS-3 solution is regulated as a drug but is not intended to provide a direct therapeutic benefit
- Arm 2 : SOLX Cold Storage: SOLX (Investigational Product)
  SOLX (Investigational): SOLX is regulated as a drug but is not intended to provide a direct therapeutic benefit.
- Arm 1: Control Room Temperature Storage/Filtration; Arm 2: Control Cold Storage: AS-3 (Control)
  AS-3 (Control): AS-3 solution is regulated as a drug but is not intended to provide a direct therapeutic benefit
Arm/Group | Arm 1: SOLX Room Temperature Storage/Filtration | Arm 2 : SOLX Cold Storage | Arm 1: Control Room Temperature Storage/Filtration | Arm 2: Control Cold Storage
Number analyzed (Participants) | 60 | 58 | 60 | 58
% recovery at day 0 | 92.57 (1.76) | 92.70 (2.34) | 90.96 (2.18) | 90.23 (3.46)

2. Primary Outcome: Residual Leukocyte Count
Description: The level of residual white blood cells in whole blood filtered after either <8 hours (AS-3) or 20-24hours (SOLX) of room temperature storage or cold storage for 72 hours.
Time Frame: <8 hours and 20-24 hours
Population: Evaluable population
Measure: Mean (Standard Deviation); unit: rWBC count (# rWBC x 10^5/unit)
Groups:
- Arm 1: SOLX Room Temperature Storage/Filtration; Arm 2 : SOLX Cold Storage: SOLX (Investigational Product)
  SOLX (Investigational): SOLX is regulated as a drug but is not intended to provide a direct therapeutic benefit.
Arm/Group | Arm 1: SOLX Room Temperature Storage/Filtration | Arm 2 : SOLX Cold Storage | Arm 1: Control Room Temperature Storage/Filtration | Arm 2: Control Cold Storage
Number analyzed (Participants) | 67 | 61 | 64 | 64
rWBC count (# rWBC x 10^5/unit) | 2.53 (2.20) | 1.25 (3.78) | 1.00 (0.45) | 0.84 (0.50)

ADVERSE EVENTS:
Time Frame: Events self-reported by the study donors were recorded within 24 hours of the completion of blood donation
Description: The investigational product (SOLX) does not come in contact with the blood donors. Therefore, all adverse events are related to standard blood donation only.
Arm/Group | Arm 1: SOLX Room Temperature Storage/Filtration | Arm 2 : SOLX Cold Storage | Arm 1: Control Room Temperature Storage/Filtration | Arm 2: Control Cold Storage
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/88 | 0/82 | 0/88
Other Adverse Events (participants affected / at risk) | 1/82 | 4/88 | 3/82 | 1/88
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: SOLX Room Temperature Storage/Filtration (N=82) | Arm 2 : SOLX Cold Storage (N=88) | Arm 1: Control Room Temperature Storage/Filtration (N=82) | Arm 2: Control Cold Storage (N=88)
Vasvagal reaction to blood donation (vascular access) (Psychiatric disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1) — Verbatim terms that fit into this category are: "Mild pallor & complaining of 'getting warm'", "Lightheadedness", "After needle inserted, donor stated they 'felt weird'", "Vasovagal syncope", "Donor was light-headed and nauseous during donation".
Hematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Refers in both cases to mild hematoma at the site of vascular access

LIMITATIONS AND CAVEATS:
The evaluable population is defined as any blood donation from which a full unit of blood was obtained. Note that the 'evaluability' status could change over time if a sample was inadvertently destroyed, overlooked or otherwise could not be analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less